CLINICAL TRIAL: NCT01470703
Title: Extracorporeal Membrane Oxygenation(ECMO) for Severe Acute Respiratory Distress Syndrome (ARDS)
Brief Title: Extracorporeal Membrane Oxygenation for Severe Acute Respiratory Distress Syndrome
Acronym: EOLIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Maquet Cardiopulmonary GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P081224; 2009-A01026-51 (Other: IDRCB)
Record Dates: First submitted 2011-11-09; First posted 2011-11-11 (Estimated); Last update posted 2018-12-21 (Actual); Status verified 2017-09

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS)
Keywords: Acute Respiratory Distress Syndrome,; ECMO, Extracorporeal Membrane Oxygenation; Randomized controlled trial; Positive-Pressure ventilation; Survival Rate
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Extracorporeal Membrane Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ECMO arm (Experimental)
  Interventions: Device: ECMO (Quadrox®, Jostra®, Maquet®)
- conventional arm (Active Comparator)
  Interventions: Other: conventional care

INTERVENTIONS:
Device: ECMO (Quadrox®, Jostra®, Maquet®) — ECMO will be initiated as rapidly as possible by venovenous access. The material to be used consists of pre-heparinized cannulae and tubing, a centrifuge pump (CardioHelp®) and a heparinized membrane oxygenator (Quadrox®, Jostra®, Maquet®). To minimize the trauma induced by mechanical ventilation, the following ventilator settings will be used: volume-assist control mode, FiO2 30-60%, PEEP ≥10 cm H2O, VT lowered to obtain a plateau pressure <25 cm H2O, respiration rate (RR) 10-30/minute or APRV mode with high pressure level <25 cm H2O and low pressure level ≥10 cm H2O
  Other Names: ECMO
  Arms: ECMO arm
Other: conventional care — Standard management of ARDS, according to the modalities applied by the 'maximal pulmonary recruitment' group in the EXPRESS trial (1): assist-controlled ventilatory mode, VT set at 6 ml/kg of ideal body weight and PEEP set so as not to exceed a plateau pressure of 28-30 cm H2O. In the case of refractory hypoxemia, the usual adjunctive therapeutics can be used: NO, prone position, HFO ventilation, almitrine infusion. A cross-over option to ECMO will be possible in the case of refractory hypoxemia defined as blood arterial saturation SaO2 <80% for >6 hours, despite mandatory use of recruitment maneuvers, and inhaled NO/prostacyclin and if technically possible a test of prone position, and only if the patient has no irreversible multiple organ failure and if the physician in charge of the patient believes that this could actually change the outcome
  Arms: conventional arm

SUMMARY:
This international multicenter, randomized, open trial will evaluate the impact of Extracorporeal Membrane Oxygenation (ECMO), instituted early after the diagnosis of acute respiratory distress syndrome (ARDS) not evolving favorably after 3-6 hours under optimal ventilatory management and maximum medical treatment, on the morbidity and mortality associated with this disease.

DETAILED DESCRIPTION:
Background: The acute respiratory distress syndrome (ARDS) is generally a severe pulmonary disease, whose associated mortality remains high. The most severe forms of ARDS, during which the hypoxemia induced by the lung involvement is the most profound, have an even more dismal prognosis, with a mortality rate exceeding 60%, despite resorting to exceptional adjunctive therapies, like NO inhalation, prone positioning of the patients, almitrine infusion or high frequency oscillation (HFO)-type ventilation. In these situations, certain teams propose establishing an extracorporeal circuit, combining a centrifuge pump and an oxygenator membrane, to assure total pulmonary assistance (oxygenation and CO2 removal from the blood), or Extra-Corporeal Membrane Oxygenation (ECMO). The aim of ECMO is to minimize the trauma induced by mechanical ventilation and to allow the lungs to rest. Unfortunately, trials evaluating ECMO for this indication over the past few decades were failures because of the interval between the onset of the disease and the installation of assistance, the poor oxygenation and CO2-removal capacities of the devices used, and the high rate of complications linked to the apparatus (massive hemorrhages resulting from intense anticoagulation and the poor 'biocompatibility' of the circuits). However, over the past few years, decisive progress has been made in the conception and construction of ECMO circuits, rendering them more 'biocompatible', better performing and more resistant. Finally, the results of the therapeutic trial (CESAR, UK) that used the latest generation ECMO are promising. Thus, the investigators now have strong clinical and pathophysiological rationales to evaluate, through a clinical trial with sufficient statistical power, the impact of early ECMO installation for the most severe forms of ARDS. This project integrates into a network (REVA or Network for Mechanical Ventilation) program.

Study hypothesis: ECMO, instituted early after the diagnosis of ARDS not evolving favorably after 3-6 hours under optimal ventilatory management and maximum medical treatment, would lower the morbidity and mortality associated with this disease.

Methods: A multicenter, randomized, open trial. Twenty-three centers will participate in this project to be conducted within the REVA network.

Experimental treatment arm: ECMO will be initiated as rapidly as possible by venovenous access. The material to be used consists of pre-heparinized cannulae and tubing, a centrifuge pump and a heparinized membrane oxygenator (Quadrox®, Jostra®, Maquet®). To minimize the trauma induced by mechanical ventilation, the following ventilator settings will be used: volume-assist control mode, FiO2 30-60%, PEEP ≥ 10 cm H2O, VT lowered to obtain a plateau pressure < 25 cm H2O, respiration rate (RR) 10-30/minute or APRV mode with high pressure level < 25 cm H2O and low pressure level ≥10 cm H2O.

Control arm treatment: Standard management of ARDS, according to the modalities applied by the 'maximal pulmonary recruitment' group in the EXPRESS trial (1): assist-controlled ventilatory mode, VT set at 6 ml/kg of ideal body weight and PEEP set so as not to exceed a plateau pressure of 28-30 cm H2O. In the case of refractory hypoxemia, the usual adjunctive therapeutics can be used: NO, prone position, HFO ventilation, almitrine infusion. A cross-over option to ECMO will be possible in the case of refractory hypoxemia defined as blood arterial saturation SaO2 < 80% for > 6 hours, despite mandatory use of recruitment maneuvers, and inhaled NO/prostacyclin and if technically possible a test of prone position, and only if the patient has no irreversible multiple organ failure and if the physician in charge of the patient believes that this could actually change the outcome.

Objective and judgement criteria: The primary endpoint is to achieve, with ECMO, significantly lower mortality on day (D) 60 (D1 is the day of randomization). Secondary objectives are to show: a benefit in terms of lower ICU and hospital mortality rates at D30 and D90; lower pneumothorax frequency; shortened duration of mechanical ventilation; less need for hemodynamic support with catecholamines; shorter ICU and hospital stays; and more days, between inclusion and D60, without mechanical ventilation, without organ failure and without hemodynamic support.

Statistical analyses: The high mortality rate of severe ARDS (≥ 60%) justifies combining all efforts to reach a rapid conclusion and thus resorting to a sequential analytical plan, with stopping rules based on the triangular test. Thus, with 80% power and a 5% α-risk for the hypothesis of ECMO achieving a 20% absolute mortality reduction, the characteristics of the study, calculated with a triangle test, are the following: a maximum of 331 subjects to be included and a 90% probability of stopping the study before 220 subjects have been included.

ELIGIBILITY:
Inclusion criteria :

1. ARDS defined according to the following criteria (9) :

   * Intubation and mechanical ventilation for ≤ 6 days
   * Bilateral radiological pulmonary infiltrates consistent with edema
   * PaO2/FiO2 ratio < 200 mm Hg
   * Absence of clinical evidence of elevated left atrial pressure and/or pulmonary arterial occlusion pressure ≤ 18 mm Hg
2. One of the 3 following criteria of disease severity:

   i. PaO2/FiO2 < 50 mm Hg with FiO2 ≥ 80% for > 3 hours, despite optimization of mechanical ventilation (Vt set at 6 ml/kg and trial of PEEP ≥ 10 cm H2O) and despite possible recourse to usual adjunctive therapies (NO, recruitment maneuvers, prone position, HFO ventilation, almitrine infusion) OR

   ii. PaO2/FiO2 < 80 mm Hg with FiO2 ≥ 80% for > 6 hours, despite optimization of mechanical ventilation (Vt set at 6 ml/kg and trial of PEEP ≥ 10 cm H2O) and despite possible recourse to usual adjunctive therapies (NO, recruitment maneuvers, prone position, HFO ventilation, almitrine infusion) OR

   iii. pH < 7.25 (with PaCO2 ≥60 mm Hg) for > 6 hours (with respiratory rate increased to 35/min) resulting from MV settings adjusted to keep plat ≤ 32 cm H2O (first, tidal volume reduction by steps of 1 mL/kg to 4 mL/kg then PEEP reduction to a minimum of 8 cm H2O.
3. Obtain informed consent from a close relative or surrogate. Should such a person be absent, the patient will be randomized according to the specifications of emergency consent and the patient will be asked to give his/her consent for the continuation of the trial when his/her condition will allow.

Exclusion criteria :

1. Intubation and mechanical ventilation for ≥ 7 days
2. Age < 18 years
3. Pregnancy
4. Weight > 1 kg/cm or BMI > 45 kg/m²
5. Chronic respiratory insufficiency treated with oxygen therapy of long duration and/or long-term respiratory assistance
6. Cardiac failure requiring veno-arterial ECMO
7. Previous history of heparin-induced thrombopenia
8. Oncohaematological disease with fatal prognosis within 5 years
9. Patient moribund on the day of randomization or has a SAPS II > 90
10. Non drug-induced coma following cardiac arrest
11. Irreversible neurological pathology, for example, flat EEG tracing cerebral herniation…
12. Decision to limit therapeutic interventions
13. ECMO cannula access to femoral vein or jugular vein impossible.
14. CardioHelp device not immediately available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2011-12-08 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
All cause mortality on day 60 following randomization | 60 days

SECONDARY OUTCOMES:
mortality on day 30 in-ICU or in-hospital mortality | 30 days
mortality on day 90 in-ICU or in-hospital mortality | 90 days
Mortality in-ICU or in-hospital mortality | at days 30, 60 and 90
  considering patients of the control group who received rescue ECMO as treatment failure (i.e. deceased on the day they received ECMO)
Mortality in-ICU or in-hospital mortality | at days 30, 60 and 90
  using a per-protocol analysis, comparing patients who received ECMO vs. others ECMO for severe ARDS

CONTACTS AND LOCATIONS:
Overall Officials: Combes Alain, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Groupe Hospitalier Pitié Salpêtrière, Paris, France

REFERENCES:
- [Background] Combes A, Hajage D, Capellier G, Demoule A, Lavoue S, Guervilly C, Da Silva D, Zafrani L, Tirot P, Veber B, Maury E, Levy B, Cohen Y, Richard C, Kalfon P, Bouadma L, Mehdaoui H, Beduneau G, Lebreton G, Brochard L, Ferguson ND, Fan E, Slutsky AS, Brodie D, Mercat A; EOLIA Trial Group, REVA, and ECMONet. Extracorporeal Membrane Oxygenation for Severe Acute Respiratory Distress Syndrome. N Engl J Med. 2018 May 24;378(21):1965-1975. doi: 10.1056/NEJMoa1800385. PMID 29791822
- [Derived] Schmidt M, Combes A. Influence of ventilatory strategy on the PRESERVE mortality risk score: response to Camporota et al. Intensive Care Med. 2014 Jun;40(6):916. doi: 10.1007/s00134-014-3284-x. Epub 2014 Apr 10. No abstract available. PMID 24718643
- [Derived] Schmidt M, Pellegrino V, Combes A, Scheinkestel C, Cooper DJ, Hodgson C. Mechanical ventilation during extracorporeal membrane oxygenation. Crit Care. 2014 Jan 21;18(1):203. doi: 10.1186/cc13702. PMID 24447458
- [Derived] Schmidt M, Zogheib E, Roze H, Repesse X, Lebreton G, Luyt CE, Trouillet JL, Brechot N, Nieszkowska A, Dupont H, Ouattara A, Leprince P, Chastre J, Combes A. The PRESERVE mortality risk score and analysis of long-term outcomes after extracorporeal membrane oxygenation for severe acute respiratory distress syndrome. Intensive Care Med. 2013 Oct;39(10):1704-13. doi: 10.1007/s00134-013-3037-2. Epub 2013 Aug 2. PMID 23907497